CLINICAL TRIAL: NCT00836745
Title: Non-Interventional Study Of Indian Patients With Advanced Renal Cell Cancer Receiving Therapy With Sutent
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181181
Record Dates: First submitted 2009-02-02; First posted 2009-02-04 (Estimated); Results first posted 2013-12-20 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-11

CONDITIONS: Renal Cell Carcinoma
Keywords: Advanced renal cell Cancer; Non interventional study; Renal Cancer; Sutent; Metastatic; Advanced Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Neoplasm Metastasis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Non Interventional
  Interventions: Other: Non Interventional

INTERVENTIONS:
Other: Non Interventional — Sutent capsule, once daily administered per the locally approved product information.
  Other Names: Observational

SUMMARY:
The Sutent® Observational Study is being proposed to assess the real-world usage patterns and effectiveness and tolerability of treatment of Indian patients with advanced renal cell cancer with Sutent®. Generation of such information is expected to aid everyday clinical decision-making by Indian doctors and will add to the body of generalizable evidence.

DETAILED DESCRIPTION:
The assignment of the patient to Sutent® treatment is not decided in advance by this noninterventional study protocol, but falls within current practice. The decision to prescribe Sutent® is clearly not driven by the decision to include the patient in this study.The sample size for this study is not based on statistical considerations. It is expected that a minimum of 100 patients will be enrolled in the study by the end of the first year and the data collected would be adequate to fulfill the observational objectives of the study.The study will be initiated at 10 sites across India during the 1st year. The study may be expanded with the addition of new sites during the 2nd year.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced renal cell cancer
* Treatment naïve or cytokine refractory

Exclusion Criteria:

* Patients presenting with a known hypersensitivity to Sunitinib or its metabolites

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with advanced renal cell cancer in the treatment naïve or cytokine refractory settings prescribed Sutent® will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2009-03; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- India (7):
  - Pfizer Investigational Site, Jaipur, Jaipur
  - Pfizer Investigational Site, Bangalore, Karnataka
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, New Delhi, National Capital Territory of Delhi
  - Pfizer Investigational Site, Chandigard, Punjab
  - Pfizer Investigational Site, Kolkata, West Bengal
  - Pfizer Investigational Site, Delhi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181181&StudyName=Non-Interventional%20Study%20Of%20Indian%20Patients%20With%20Advanced%20Renal%20Cell%20Cancer%20Receiving%20Therapy%20With%20Sutent

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: Participants who received sunitinib capsule once daily as per local product information, were followed up for 1 year or till the occurrence of disease progression, early discontinuation of sunitinib therapy (due to unacceptable toxicity, participant's request or lost to follow up), or death, whichever occurred earlier. Sunitinib dose was adjusted solely according to medical and therapeutic needs.
Period: Overall Study
Arm/Group | Sunitinib
Started | 36
Completed | 15
Not Completed | 21
Not completed — Death | 2
Not completed — Lost to Follow-up | 10
Not completed — Adverse Event | 3
Not completed — Objective progression or relapse | 4
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS defined as the time (in weeks) from the date of first dose of sunitinib to the date of first documentation of objective tumor progression or death due to any cause, whichever occurs first. Date of first documentation of progression was based on radiological assessment of tumor measurements. PFS was calculated as (first event date minus the date of first dose of study medication plus 1) divided by 7.
Time Frame: Baseline until disease progression or death due to any cause or discontinuation from study treatment (up to 1 year from start of first dose)
Population: Data was not analyzed since PFS for all participants was censored either due to inadequate baseline assessments, absence of on-study disease assessment, or being on follow-up for progression.
Arm/Group | Sunitinib
Number analyzed (Participants) | 0

2. Secondary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to response evaluation criteria in solid tumors (RECIST). Confirmed responses were those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR defined as the disappearance of all lesions (target and/or non- target). PR those with at least 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline until disease progression or discontinuation from study treatment (up to 1 year from start of first dose)
Population: Per protocol (PP) analysis set included all enrolled participants who had the disease under study, measurable disease and an adequate baseline disease assessment, and who started sunitinib treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 4
percentage of participants | 0 [0.0 to 60.2]

3. Secondary Outcome: Number of Participants Who Required Management of Skin and Subcutaneous Tissue Related Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Number of participants who required dose modifications and other measures for the management of skin and subcutaneous tissue related adverse events were presented.
Time Frame: Baseline up to 1 year from start of first dose
Population: Safety analysis set included all enrolled participants who started treatment with sunitinib.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 36
participants
  Dose Reduction | 1
  Dose Interruption | 1
  Avoidance of Hot water for Cleaning Hands and Feet | 1

4. Secondary Outcome: Number of Participants Who Required Management of Other Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Number of participants who required dose modifications and other measures for the management of other adverse events were to be presented.
Time Frame: Baseline up to 1 year from start of first dose
Population: Safety analysis set included all enrolled participants who started treatment with sunitinib.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 36
participants | 20

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 7/36
Other Adverse Events (participants affected / at risk) | 20/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=36)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiopulmonary failure (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Disease progression (General disorders) | 1
Diabetic foot infection (Infections and infestations) | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 1
Haematuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=36)
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Odynophagia (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Adverse event (General disorders) | 1
Asthenia (General disorders) | 3
Chills (General disorders) | 1
Fatigue (General disorders) | 1
Mucosal inflammation (General disorders) | 2
Oedema (General disorders) | 2
Pyrexia (General disorders) | 3
Cholelithiasis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 4
Abdominal wall abscess (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Alanine aminotransferase (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase (Investigations) | 3
Aspartate aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase (Investigations) | 2
Blood creatinine (Investigations) | 2
Blood lactate dehydrogenase (Investigations) | 1
Neutrophil count (Investigations) | 1
Platelet count (Investigations) | 1
Weight decreased (Investigations) | 4
Weight increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Investigations) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Bladder spasm (Renal and urinary disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Relatively small sample size might limit any useful interpretation and applicability of data for larger populations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.